CLINICAL TRIAL: NCT00124267
Title: Efficacy of Intrarectal Versus Intravenous Quinine for the Treatment of Childhood Cerebral Malaria: a Randomized Clinical Trial
Brief Title: Efficacy of Intrarectal Versus Intravenous Quinine for the Treatment of Childhood Cerebral Malaria
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Makerere University (Other)
Collaborators: Sanofi-Synthelabo (Industry); Ministry of Health, Uganda (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2001/HD11/524/RQ
Record Dates: First submitted 2005-07-26; First posted 2005-07-27 (Estimated); Last update posted 2005-08-04 (Estimated); Status verified 2005-07

CONDITIONS: Cerebral Malaria
Keywords: Cerebral; malaria; intra-rectal; quinine; children; Uganda; efficacy; safety
MeSH Terms: conditions — Malaria, Cerebral; Malaria

INTERVENTIONS:
Drug: Intrarectal quinine

SUMMARY:
Cerebral malaria is the most lethal complication of P.falciparum infection with a mortality rate between 5 and 40%. Intravenous quinine remains the recommended treatment for cerebral malaria. However its administration is often not feasible due to lack of simple equipment or trained staff. When referral is not possible, a viable alternative is needed. The intrarectal route is of interest in children since it is painless and simple. Studies of the efficacy of intrarectal quinine in the treatment of cerebral malaria are limited. The study aims to establish the efficacy of intrarectal quinine in the treatment of childhood cerebral malaria.

DETAILED DESCRIPTION:
Cerebral malaria is the most lethal complication of P.falciparum infection with a mortality rate between 5 and 40%. Intravenous quinine remains the recommended treatment for cerebral malaria. However its administration is often not feasible due to lack of simple equipment or trained staff. When referral is not possible, a viable alternative is needed. The intrarectal route is of interest in children since it is painless and simple. A few studies in Francophone Africa have reported clinical efficacy and tolerance of intrarectal quinine. Although the studies were randomized trials, they were not blinded and did not use the WHO definition of cerebral malaria as selection criteria.

The current study aims to establish whether intrarectal quinine is as effective and as safe as intravenous quinine in the treatment of childhood cerebral malaria.

To address the shortcomings of the Francophone African studies, the investigators have designed a randomized, double blind placebo controlled clinical trial to include patients who meet the WHO definition of cerebral malaria.

Hypothesis:

Intrarectal quinine (15mg/kg every 8 hours) given to children with cerebral malaria, will lead to a shorter parasite clearance time (39.9 hours) than intravenous quinine (55.0 hours).

The investigators calculated a sample size of 54 patients in each group for 90% power and 95% confidence. In the calculation, the researchers assumed that the children receiving intrarectal quinine would have a mean parasite clearance time of 39.9 (SD 24.3) hours and those receiving intravenous quinine would have a mean parasite clearance time of 55.0(SD 24.3) hours (27.5% effect size), according to a study by Aceng, Byarugaba and Tumwine in the same hospital.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to 5 years admitted to Mulago hospital during the study period who satisfy the World Health Organization (WHO) case definition of cerebral malaria (Unarousable coma lasting more than 30 minutes after a seizure, with peripheral asexual P.falciparum parasitaemia and absence of other causes of coma) and whose caretakers give informed consent.

Exclusion Criteria:

* Patients with diarrhea (more than 4 motions/24 hours)
* Any recent anal pathology (such as rectal bleeding, rectal prolapse)
* Documented quinine treatment in previous 48 hours.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108
Dates: Start 2003-09; Study Completion 2004-01

PRIMARY OUTCOMES:
Parasite clearance time

SECONDARY OUTCOMES:
Fever clearance time
Coma recovery time
Time to sit unsupported
Time to begin oral intake
Mortality
Neurological sequelae
Adverse drug events

CONTACTS AND LOCATIONS:
Overall Officials: Jane Achan, MBChB, Principal Investigator — Department of Paediatrics and Child Health, Makerere University
Locations (1):
- Mulago Hospital, Kampala, Kampala, Uganda

REFERENCES:
- [Background] Pussard E, Straczek C, Kabore I, Bicaba A, Balima-Koussoube T, Bouree P, Barennes H. Dose-dependent resorption of quinine after intrarectal administration to children with moderate Plasmodium falciparum malaria. Antimicrob Agents Chemother. 2004 Nov;48(11):4422-6. doi: 10.1128/AAC.48.11.4422-4426.2004. PMID 15504872
- [Background] Barennes H, Sterlingot H, Nagot N, Meda H, Kabore M, Sanou M, Nacro B, Bouree P, Pussard E. Intrarectal pharmacokinetics of two formulations of quinine in children with falciparum malaria. Eur J Clin Pharmacol. 2003 Feb;58(10):649-52. doi: 10.1007/s00228-002-0546-2. Epub 2003 Jan 29. PMID 12610739
- [Background] Barennes H, Munjakazi J, Verdier F, Clavier F, Pussard E. An open randomized clinical study of intrarectal versus infused Quinimax for the treatment of childhood cerebral malaria in Niger. Trans R Soc Trop Med Hyg. 1998 Jul-Aug;92(4):437-40. doi: 10.1016/s0035-9203(98)91083-5. PMID 9850403
- [Background] Aceng JR, Byarugaba JS, Tumwine JK. Rectal artemether versus intravenous quinine for the treatment of cerebral malaria in children in Uganda: randomised clinical trial. BMJ. 2005 Feb 12;330(7487):334. doi: 10.1136/bmj.330.7487.334. PMID 15705690
- [Background] Simoes EA, Peterson S, Gamatie Y, Kisanga FS, Mukasa G, Nsungwa-Sabiiti J, Were MW, Weber MW. Management of severely ill children at first-level health facilities in sub-Saharan Africa when referral is difficult. Bull World Health Organ. 2003;81(7):522-31. Epub 2003 Sep 3. PMID 12973645
- [Derived] Nakibuuka V, Ndeezi G, Nakiboneka D, Ndugwa CM, Tumwine JK. Presumptive treatment with sulphadoxine-pyrimethamine versus weekly chloroquine for malaria prophylaxis in children with sickle cell anaemia in Uganda: a randomized controlled trial. Malar J. 2009 Oct 24;8:237. doi: 10.1186/1475-2875-8-237. PMID 19852829